CLINICAL TRIAL: NCT03429790
Title: A Randomised Controlled Trial of Intra-Operative Cell Salvage During Caesarean Section in Women Needing Blood Transfusion
Brief Title: Cell Salvage During Caesarean Section (CSCS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The staff of the research team changed and it was impossible to continue, so it was terminated
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Ting Li, associate chief physician, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSCS
Record Dates: First submitted 2017-06-25; First posted 2018-02-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Blood Transfusion
Keywords: caesarean section; cell salvage; blood transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group intra-operative cell salvage (Experimental): The theoretical amount of blood transfusion should be based on the following formula:
  The amount of blood transfusion needed (ML) * Hb= (Hb2-Hb1) * blood volume of blood transfusion Hb1: actual measured hemoglobin; Hb2: target hemoglobin (100 g / L) Blood volume = 100ml/kg * body weight The difference between the actual blood transfusion and the theoretical blood transfusion should be controlled within ± 15% of the theoretical blood transfusion (in terms of hemoglobin), whether the experimental group or the no intervention group.
  Interventions: Combination Product: intra-operative cell salvage; Combination Product: allogeneic blood transfusion
- group allogeneic blood transfusion (Active Comparator): The theoretical amount of blood transfusion should be based on the following formula:
  The amount of blood transfusion needed (ML) * Hb= (Hb2-Hb1) * blood volume of blood transfusion Hb1: actual measured hemoglobin; Hb2: target hemoglobin (100 g / L) Blood volume = 100ml/kg * body weight The difference between the actual blood transfusion and the theoretical blood transfusion should be controlled within ± 15% of the theoretical blood transfusion (in terms of hemoglobin), whether group intra-operative cell salvage or group allogeneic blood transfusion.
  Interventions: Combination Product: allogeneic blood transfusion

INTERVENTIONS:
Combination Product: intra-operative cell salvage — intra-operative cell salvage collects the patient's blood lost during an operation, processes it and returns it to their own circulation.
  Arms: group intra-operative cell salvage
Combination Product: allogeneic blood transfusion — transfuse allogeneic blood to patients if blood transfusion is needed.

SUMMARY:
The purposes of this study are:

1. To compare the difference of blood loss of the patients undergoing cesarean section between intraoperative blood recovery and allogeneic blood transfusion.
2. To compare the safety of the two methods.
3. To evaluate the medical cost and the overall cost of the two methods.

DETAILED DESCRIPTION:
Preoperative: 1.To select patients according to the criteria.2.To obtain the consent of the obstetrician, the anesthesiologist, and the patients.

Intraoperative:According to local blood transfusion guidelines, obstetric advice, anesthesia advice(tentative: before a blood transfusion maternal's Hb less than 70g/L or Hb:70-100g/l before a blood transfusion according to the blood transfusion program and doctor's determine to do the blood transfusion),those who need blood transfusion during cesarean section will be randomly assigned to the following two groups:

1. cesarean section using intraoperative blood recovery group (test group).
2. cesarean section using allogeneic blood transfusion group (control group).

The theoretical amount of blood transfusion should be based on the following formula:

The amount of blood transfusion needed (ML) * Hb= (Hb2-Hb1) * blood volume of blood transfusion Hb1: actual measured hemoglobin; Hb2: target hemoglobin (100 g / L) Blood volume = 100ml/kg * body weight The difference between the actual blood transfusion and the theoretical blood transfusion should be controlled within ± 15% of the theoretical blood transfusion (in terms of hemoglobin), whether the test group or the control group.

Postoperative: Calculate the amount of bleeding in the subjects and other related indicators.

Follow up: maternal pregnancy again: detection of maternal blood group antibody IgG titer, hemolytic disease of the newborn Statistical data: the specially assigned person is responsible for the data collection. And the data is entryed by two times (the first phase: hospitalization period, the second phase: follow-up), which is by the inspectors to verify the authenticity and traceability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Delivery by elective or emergency caesarean section with an identifiable increased risk of haemorrhage.
* Ability to provide informed consent
* Participants need blood transfusion

Exclusion Criteria:

* Hb<70g/L before operation
* Participants have a history of blood transfusion
* Blood type is RH blood type
* Sickle cell disease
* The obstetricians and anesthesia doctors think some cases existing intraoperatie blood recycling contraindications
* PT and APTT is 1.5 times longer than normal and above, or platelet is less than 50 * 109 / L preoperative
* Cultural or social beliefs contraindicating blood transfusion.
* Significant antibodies making it difficult to find cross matched blood for transfusion
* participation in another clinical trial within 3 months prior to selection
* ability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
blood loss of the subjects in 5 days of after operation | in fifth day post operation
  calculate the changes of Hct and the amount of blood transfusion

SECONDARY OUTCOMES:
postoperative Hct in first day post operation | in first day post operation
  the Hct in first day post operation
postoperative Hb in first day post operation | in first day post operation
  the Hb in first day post operation
postoperative PT in first day post operation | in first day post operation
  the PT in first day post operation
postoperative APTT in first day post operation | in first day post operation
  the APTT in first day post operation
postoperative Hct in the fifth day post operation | in the fifth day post operation
  the Hct in fifth day post operation
postoperative Hb in the fifth day post operation | in the fifth day post operation
  the Hb in fifth day post operation
postoperative PT in the fifth day post operation | in the fifth day post operation
  the PT in fifth day post operation
postoperative APTT in the fifth day post operation | in the fifth day post operation
  the APTT in fifth day post operation
Total intraoperative and postoperative blood transfusion | from the date of operation until the date of hospital discharge, assessed up to 7 days
  calculate the amount of blood transfusion
Length of hospital stay | from the date of operation until the date of hospital discharge, assessed up to 7 days
  calculate the length of hospital stay
first mobilization | from the date of operation up to first mobilization, assessed up to 7 days
  calculate the time to first mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Fang Gao Smith, M.D., Study Chair — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Qingquan Lian, M.D., Study Chair — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Ting LI, M.D., Principal Investigator — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University

REFERENCES:
- [Background] Cantwell R, Clutton-Brock T, Cooper G, Dawson A, Drife J, Garrod D, Harper A, Hulbert D, Lucas S, McClure J, Millward-Sadler H, Neilson J, Nelson-Piercy C, Norman J, O'Herlihy C, Oates M, Shakespeare J, de Swiet M, Williamson C, Beale V, Knight M, Lennox C, Miller A, Parmar D, Rogers J, Springett A. Saving Mothers' Lives: Reviewing maternal deaths to make motherhood safer: 2006-2008. The Eighth Report of the Confidential Enquiries into Maternal Deaths in the United Kingdom. BJOG. 2011 Mar;118(Suppl 1):1-203. doi: 10.1111/j.1471-0528.2010.02847.x. PMID 21356004
- [Background] Bodelon C, Bernabe-Ortiz A, Schiff MA, Reed SD. Factors associated with peripartum hysterectomy. Obstet Gynecol. 2009 Jul;114(1):115-123. doi: 10.1097/AOG.0b013e3181a81cdd. PMID 19546767
- [Background] Waters JH, Biscotti C, Potter PS, Phillipson E. Amniotic fluid removal during cell salvage in the cesarean section patient. Anesthesiology. 2000 Jun;92(6):1531-6. doi: 10.1097/00000542-200006000-00008. PMID 10839901
- [Background] Sullivan I, Faulds J, Ralph C. Contamination of salvaged maternal blood by amniotic fluid and fetal red cells during elective Caesarean section. Br J Anaesth. 2008 Aug;101(2):225-9. doi: 10.1093/bja/aen135. Epub 2008 May 30. PMID 18515817
- [Background] Catling S. Intraoperative cell salvage in obstetrics. Clin Risk 2008 Jan 1;14(1):14-7.
- [Background] Zheng J, Du L, Du G, Liu B. Coagulopathy associated with cell salvage transfusion following cerebrovascular surgery. Pak J Med Sci. 2013 Nov;29(6):1459-61. doi: 10.12669/pjms.296.3750. PMID 24550976
- [Background] Sullivan IJ, Hicks MK, Faulds JN, Carson PJ, Noble RS. A modified thrombin clotting time test as a quality control marker for heparin contamination in obstetric intraoperative cell salvage. Transfus Med. 2012 Feb;22(1):68-70. doi: 10.1111/j.1365-3148.2011.01123.x. Epub 2011 Dec 16. PMID 22171556
- [Background] Elagamy A, Abdelaziz A, Ellaithy M. The use of cell salvage in women undergoing cesarean hysterectomy for abnormal placentation. Int J Obstet Anesth. 2013 Nov;22(4):289-93. doi: 10.1016/j.ijoa.2013.05.007. Epub 2013 Aug 16. PMID 23958277
- [Background] Jansen AJ, van Rhenen DJ, Steegers EA, Duvekot JJ. Postpartum hemorrhage and transfusion of blood and blood components. Obstet Gynecol Surv. 2005 Oct;60(10):663-71. doi: 10.1097/01.ogx.0000180909.31293.cf. PMID 16186783

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03429790/Prot_SAP_ICF_000.pdf